CLINICAL TRIAL: NCT01732302
Title: Educational Intervention to Reduce Drug-related Hospitalizations and Visits in Emergency Departments in Elderly Primary Health Care Patients - a Cluster-randomized Controlled Trial
Brief Title: Educational Intervention to Reduce Drug-related Hospitalizations in Elderly Primary Health Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Lars Agreus, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012 1266-31
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Polypharmacy; Adverse Drug Reaction
Keywords: Drug Utilization Review; Aged; Aged, 80 and over; Primary Health Care
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational intervention (Experimental): Primary health care centers (PHCC) in the intervention group will be visited twice by a pharmacist within a period of three months. At the first visit, an educational intervention will focus on two properties: on the one hand, feed-back of actual patient data of the PHCC illustrating the primary-health-care-specific characteristics of inappropriate prescribing in the elderly patient will be given. Education of relevant subjects will be given in relation to detected problems. On the other hand, a clinical routine regarding the performance of drug utilization reviews will be developed in cooperation with the health care providers. At the second visit 3 months later, the developed concept will be critically reviewed and eventually developed further.
  Interventions: Other: Educational intervention
- Delayed educational intervention (No Intervention): Primary health care centers in the delayed intervention group will receive the same intervention as described above with 9 months delay.

INTERVENTIONS:
Other: Educational intervention — Primary health care centers (PHCC) in the intervention group will be visited twice by a pharmacist within a period of three months. At the first visit, an educational intervention will focus on two properties: on the one hand, feed-back of actual patient data of the PHCC illustrating the primary-health-care-specific characteristics of inappropriate prescribing in the elderly patient will be given. Education of relevant subjects will be given in relation to detected problems. On the other hand, a clinical routine regarding the performance of drug utilization reviews will be developed in cooperation with the health care providers. At the second visit 3 months later, the developed concept will be critically reviewed and eventually developed further.
  Arms: Educational intervention

SUMMARY:
The purpose of this study is to determine whether an educational intervention given towards health care providers working in primary health care centers can reduce inappropriate prescribing in the elderly patient and thus reduce number and length of drug-related hospitalizations as well as number of emergency department visits in this patient group.

DETAILED DESCRIPTION:
Inappropriate medication in the elderly patient leads to substantial morbidity, possibly causing up to 20% of hospitalizations in this patient group (1). To improve prescribing and thus reduce undesired drug effects is a great challenge for doctors and nurses in primary health care.

Performance of drug utilization reviews is recommended in order to reduce the negative impact of inappropriate prescribing in the elderly. However, scientific evidence on their efficacy is lacking, especially regarding patient-related health outcomes (2,3). Most studies are carried out in inpatient care, making it difficult to draw conclusions regarding primary health care (2). Moreover, studies in this scientific field diverge regarding the content and structure of drug utilization reviews, which implies that comparison between studies becomes challenging, if not impossible.

This trial aims at educating health care providers in how to perform drug utilization reviews, and to help them implement theory into practice.

ELIGIBILITY:
Inclusion Criteria:

* primary health care center in Stockholm County
* authorized by Stockholm County Council since at least 3 years
* at least 5% of patients attributed to primary health care center are 65 years and older
* primary health care center takes care of at least 10 home care patients

Exclusion Criteria:

* less than 3000 patients listed in primary health care center
* primary health care centers where researchers carrying out the present study work

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Composite outcome: Unplanned hospitalisation or emergency department visit | 9 months

SECONDARY OUTCOMES:
Unplanned hospitalisation | 9 months
Emergency department visit | 9 months
Length of hospital stay | 9 months
All cause mortality | 9 months
Number of drug utilization reviews | 9 months
Number of patients with polypharmacy | 9 months
  polypharmacy: 5-9 drugs/patient excessive polypharmacy: 10 and more drugs/patient
Inappropriate drug use according to national guidelines | 9 months
  see link
Number of patients with contraindicated drugs regarding renal function | 9 months
Number of drugs with inappropriate drug dose regarding renal function | 9 months
Number of drug interactions | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hasselström, MD, PhD, Principal Investigator — Centre for Family Medicine, Dept of Neurobiology, Care sciences and Society, Karolinska Institutet
Locations (1):
- Centre for Family Medicine, Dept of Neurobiology, Care sciences and Society, Karolinska Institutet, Huddinge, Sweden

REFERENCES:
- [Background] Beijer HJ, de Blaey CJ. Hospitalisations caused by adverse drug reactions (ADR): a meta-analysis of observational studies. Pharm World Sci. 2002 Apr;24(2):46-54. doi: 10.1023/a:1015570104121. PMID 12061133
- [Background] Spinewine A, Schmader KE, Barber N, Hughes C, Lapane KL, Swine C, Hanlon JT. Appropriate prescribing in elderly people: how well can it be measured and optimised? Lancet. 2007 Jul 14;370(9582):173-184. doi: 10.1016/S0140-6736(07)61091-5. PMID 17630041
- [Background] Stewart S, Pearson S, Luke CG, Horowitz JD. Effects of home-based intervention on unplanned readmissions and out-of-hospital deaths. J Am Geriatr Soc. 1998 Feb;46(2):174-80. doi: 10.1111/j.1532-5415.1998.tb02535.x. PMID 9475445